CLINICAL TRIAL: NCT06940817
Title: Re-establishing Inter-generational Cooking Education and Improving Diet Quality Through an Integrated Parenting and Healthy Cooking Program for Low-income Families With Young Children
Brief Title: Cooking HEalthy and Facilitating Early Childhood Development: CHEF-ED Study
Acronym: CHEF-ED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Sheryl Hughes, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-53855; 2023-68015-40967 (Other Grant/Funding Number: USDA NIFA)
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Teaching Healthy Cooking Skills to Parents and Their Preschool Children
Keywords: Food security; Nutrition education; Cooking practices; Feeding practices; Chronic disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CHEF-ED + Food Delivery group (Experimental): Participants in this arm will receive a one-time delivery of non-perishable basic culinary ingredients and kitchen utensils and access to the CHEF-ED program, which includes weekly online program materials, such as videos, infographics, and recipes sent via text or email over 7 weeks.
  Interventions: Behavioral: CHEF-ED + Food Delivery
- Food Delivery Only group (Active Comparator): Participants in this arm receive a one-time delivery of non-perishable basic culinary ingredients and kitchen utensils but will not have access to the CHEF-ED program during the study period.
  Interventions: Behavioral: Food Delivery Only
- Control group (No Intervention): Participants in this arm will not receive the healthy cooking ingredients delivery nor will they have access to the CHEF-ED program during the study period.

INTERVENTIONS:
Behavioral: CHEF-ED + Food Delivery — CHEF-ED is a 7-week, digital, video-based parental intervention that teaches healthy cooking practices and an optimal way to involve children in home cooking. Each week features a video, infographics, and recipe content. The content is designed to be integrated into the home food environment without major changes to shopping habits. However, some basic culinary ingredients that are featured may not already be part of participating family pantry stocks. To support participants in effectively learning the healthy cooking strategies, participating families are provided a one-time home food delivery of non-perishable basic culinary ingredients and kitchen utensils, such as cooking oil, spices, whole wheat pasta, low sodium soy sauce, bowls.
  Arms: CHEF-ED + Food Delivery group
Behavioral: Food Delivery Only — The Food Delivery Only intervention involves participants receiving a one-time home food delivery of non-perishable basic culinary ingredients and kitchen utensils, such as cooking oil, spices, whole wheat pasta, low sodium soy sauce, bowls.
  Arms: Food Delivery Only group

SUMMARY:
This study aims to test a new online program we developed for parents and their preschool children, called CHEF-ED. CHEF-ED focuses on healthy cooking, parental feeding practices, and involving children in home food preparation.

DETAILED DESCRIPTION:
All study activities take place online over a 3-month period, and participants are randomly assigned to one of three groups: the CHEF-ED + Food Delivery group, the Food Delivery Only group, or the control group. Participants will not know to which group they are assigned until after they complete the time point 1 surveys. The assignment will be determined randomly using a computer program (equivalent to flipping a coin).

To test how well the program works, regardless of group assignment, participants are asked to complete surveys at two different time points: Time point 1 = pre-program, shortly after enrollment, and Time point 2 = post-program, about 8-10 weeks later. The surveys take about 2 hours to complete online at each time point and will include questions about the participant's and their child's dietary intake, their cooking frequency/quality, food parenting practices, and program content retention. Surveys will also include questions about family's demographics (such as participant's and their child's date of birth, ethnicity, race, sex, etc.), and household food access.

The CHEF-ED + Food Delivery group receives a one-time home food delivery of healthy cooking ingredients and kitchen utensils, such as cooking oil, spices, whole wheat pasta, low sodium soy sauce, bowls, and recipe books. Participants in this group also receive links to weekly CHEF-ED online lessons via text /email message for 7 weeks. Each weekly lesson will include a short video, infographics, and recipes.

The Food Delivery Only group receives a one-time home food delivery of healthy cooking ingredients and kitchen utensils, but no other program materials.

The control group receives no program materials or food delivery.

About 8-10 weeks after completing the time point 1 surveys, participants will receive links to complete the time point 2 surveys. After completing the post-program surveys, participants who were in the Food Delivery Only or control group will receive additional program materials that were not previously provided due to their group assignment. This means that the Food Delivery Only group, after completing the time point 2 surveys, will receive links to all of the CHEF-ED program materials (videos, infographics, recipes) and, the control group, after completing the time point 2 surveys, will receive the one-time healthy ingredients and kitchen utensils delivery and links to all of the CHEF-ED program materials.

Additionally, participants in the CHEF-ED + Food Delivery group, after the post-program surveys, may be invited to take part in an interview to share their experience with the program. This interview will be conducted over the phone or a video conference platform. The information participants share during the interview, such as suggestions and insights on materials accessibility, will help us improve the program.

ELIGIBILITY:
Inclusion Criteria:

* Parents/caregivers of preschooler children ages 3 to 5 living in the greater Houston area.
* Must have access to the Internet through a smartphone, tablet, laptop, or desktop computer.
* Should be able to read, write, and communicate in English or Spanish.

Exclusion Criteria:

* Parents/caregivers and children who have any kind of food allergies, medical conditions, or dietary restrictions that may affect participation in the program.
* Parents/caregivers under the age of 18.
* Parents/caregivers of children with severe developmental delays.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Child diet quality | From baseline assessment to the post-intervention assessment. The intervention program is 7 weeks.
  Parent report of child dietary intake using a validated food frequency survey.

SECONDARY OUTCOMES:
Parent diet quality | From baseline assessment to the post-intervention assessment. The intervention program is 7 weeks.
  Self-report of diet quality using a validated diet history questionnaire.
Parent cooking frequency/quality | From baseline assessment to the post-intervention assessment. The intervention program is 7 weeks.
  Self-report of healthy cooking using a validated questionnaire.
Food parenting practices | From baseline assessment to the post-intervention assessment. The intervention program is 7 weeks.
  Second order constructs from a validated food parenting questionnaire - encourage trying new foods; structure; external control.
Knowledge of best feeding practices | From baseline assessment to the post-intervention assessment. The intervention program is 7 weeks.
  Six items related to child eating behaviors reported by parents.

OTHER OUTCOMES:
Sample characteristics | From baseline assessment to the post-intervention assessment. The intervention program is 7 weeks.
  Self-report of demographic information, food security status, and acculturation.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O. Hughes, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided